CLINICAL TRIAL: NCT06230770
Title: The Impact of Progestin-only Contraception on Bleeding Patterns in Individuals Initiating Testosterone Therapy for Gender Affirmation
Brief Title: Impact of Progestin-only Contraception on Bleeding Patterns in Individuals Initiating GATT
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sarah Averbach, MD MAS, Associate Professor, University of California, San Diego
Other Study IDs: 809057
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Gender; Contraception
Keywords: progestin; testosterone; gender-affirming; bleeding
MeSH Terms: conditions — Coitus; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Bleeding data — Participants will report their daily bleeding patterns

SUMMARY:
Gender diverse individuals who use gender-affirming testosterone therapy (GATT) to reduce gender dysphoria may also use progestins for contraception and to manage or suppress uterine bleeding. Research is limited, however, regarding expected bleeding patterns for individuals who choose to initiate GATT concurrently with a progestin. Clinicians who prescribe GATT do not have sufficient data to adequately counsel patients on side effects of concurrent progestin use and therefore extrapolate from studies conducted in cisgender women. This study is a prospective cohort study evaluating bleeding patterns and satisfaction among patients initiating GATT with or without concurrent initiation of a progestin contraceptive. The results from this study will enable clinicians to more accurately counsel patients using GATT on how the use of a progestin might affect their bleeding and whether this differs by progestin method.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking currently have a uterus and ovaries
* desire to initiate GATT
* potential desire to initiate a progestin (within 14 days of GATT initiation)

Exclusion Criteria:

* previous gender-affirming surgery to remove their uterus and/or ovaries

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will enroll 160 participants who are English-speaking, at least 18 years old, currently have a uterus and ovaries, desire to initiate GATT, and potentially desire to initiate a progestin (within 14 days of GATT initiation). To ensure generalizability of results, participants with baseline irregular bleeding will not be excluded.
  Participants who have recently initiated a progestin may be eligible for inclusion. Participants who have had gender-affirming surgery to remove their uterus and/or ovaries will not be eligible for inclusion.
  We will recruit participants from clinics in San Diego that prescribe GATT, including the UCSD OBGYN clinic, two UCSD Gender Health program affiliated clinics, and UCSD Student Health Services.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean days bleeding or spotting | Start of GATT to 30 days
  mean number of days of bleeding or spotting during the 30 days after GATT initiation

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Loeliger, MD. PhD, Study Director — UC San Diego; Sarah Averbach, MD, MSc, Principal Investigator — UC San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No